CLINICAL TRIAL: NCT01537718
Title: Evaluation of the Performances of the Sleep Disordered Breathing Monitoring Function in Pacemaker
Acronym: DREAM
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LivaNova (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IBSY04
Record Dates: First submitted 2012-02-17; First posted 2012-02-23 (Estimated); Last update posted 2013-07-17 (Estimated); Status verified 2013-07

CONDITIONS: Bradycardia
MeSH Terms: conditions — Bradycardia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- REPLY 200 implanted patients (Experimental): REPLY 200 implanted patients
  Interventions: Device: REPLY 200

INTERVENTIONS:
Device: REPLY 200 — REPLY 200 pacemaker

SUMMARY:
The IBSY04 clinical investigation is an European, prospective, multi-centre, non-randomized, longitudinal study.

DETAILED DESCRIPTION:
The purpose of this study is to assess the performance of Sleep Disordered Breathing Monitoring function (SDB) in pacemakers by comparing device diagnostic data to the results of in-lab PolySomnoGraphy (PSG) recording during the same night

ELIGIBILITY:
Inclusion Criteria: Any patient enrolled in the study must fulfil all of the following criteria:

* Patients eligible for implantation of a single or dual-chamber pacemaker according to current available guidelines
* Patients who are scheduled for implant of a REPLY 200 SR; or REPLY 200 DR pacemaker
* Patients who provide signed and dated informed consent

Exclusion Criteria:

* Inability to understand the purpose of the study or refusal to co-operate
* Unavailability for scheduled follow-ups at the implanting centre
* Already included in another clinical study that could affect the results of this study
* Inability or refusal to provide informed consent
* Patient is minor (less than 18-years old)
* Patient is pregnant (women of childbearing potential should have a negative pregnancy test prior to enrolment)
* Patient is forfeiture of freedom or under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-03; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Event-based sensitivity of breathing troubles | 1 day
  Evaluation of this outcome requires measuring the number of ventilation pauses and ventilation reductions detected during the same night using SDB Monitoring function or the reference in-lab PSG (clinical assessment).
Event-based Positive Predictive Value of breathing troubles | 1 day
  The Event-based Positive Predictive Value (PPV)of breathing troubles is complementary to Sensitivity. It is the proportion of abnormal events appropriately detected by SDB Monitoring function compared to the total number of abnormal events detected by SDB Monitoring function.

SECONDARY OUTCOMES:
Apnea Index-based Positive Predictive Value | 1 day
  The objective is to assess the Positive Prédictive Value of the SDB Monitoring function based on RDI stored in the pacemaker and the AHI derived from in-lab Polysomnography during the same night.
Apnea Index-based Negative Predictive Value | 1 day
  The objective is to assess the NPV of the SDB Monitoring function based on RDI stored in the pacemaker or the AHI derived from in-lab Polysomnography during the same night.
Safety based on Adverse events | 3 months
  The objective will allow to assess the safety with the summarize all adverse events through 3-month follow-up related to the implant procedure and pacing system or related to any other cause.

CONTACTS AND LOCATIONS:
Overall Officials: PASCAL DEFAYE, Dr, Principal Investigator — CHU Grenoble, France
Locations (5):
- France (3):
  - Créteil
  - Grenoble
  - La Rochelle
- Spain (2):
  - Barcelona
  - Seville